CLINICAL TRIAL: NCT01084187
Title: Correlation of Flow Mediated Dilation of Brachial Artery and Carotid Intima Media Thickness With Erectile Dysfunction Severity and Clinical Response to PDE 5 Inhibitor in Hypertensive Men
Brief Title: Correlation Study of Vascular Parameters in Hypertensive Men With Erectile Dysfunction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitario Pedro Ernesto (Other)
Responsible Party: Valter Javaroni, Hospital Universitário Pedro Ernesto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EDAH2010
Record Dates: First submitted 2010-03-09; First posted 2010-03-10 (Estimated); Last update posted 2011-04-18 (Estimated); Status verified 2011-04

CONDITIONS: Erectile Dysfunction; Arterial Hypertension; Endothelial Dysfunction
Keywords: erectile dysfunction; arterial hypertension; flow mediated vasodilation; endothelial dysfunction; carotid intima media thickness; vardenafil
MeSH Terms: conditions — Erectile Dysfunction; Hypertension | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- vardenafil on demand (Active Comparator): four sexual attempts with 20 mg vardenafil during next four weeks
  Interventions: Drug: Vardenafil
- placebo (Placebo Comparator): placebo of vardenafil during four weeks
  Interventions: Drug: Vardenafil
- daily vardenafil (Active Comparator): 10 mg of vardenafil each day during four weeks
  Interventions: Drug: Vardenafil

INTERVENTIONS:
Drug: Vardenafil — vardenafil 20 mg on demand or vardenafil daily or placebo
  Other Names: Levitra

SUMMARY:
The purpose of the study is to assess the correlation of FMD of brachial artery and carotid intima media thickness with ED severity and clinical response to vardenafil in hypertensive men.

DETAILED DESCRIPTION:
To achieve this objective, a prospective study will be conducted, with hypertensive patients ranging from 50 to 70 years, presenting vasculogenic erectile dysfunction for over six months and sexually actives. All patients will be assessed for clinical and laboratorial data, endothelial dysfunction, endothelium independent vasodilation and carotid intima media thickness at the inclusion of the study. They will receive medical orientations from the same urologist and will return after four attempts with 20 mg of vardenafil.

ELIGIBILITY:
Inclusion Criteria:

* arterial hypertension and erectile dysfunction of vascular origin for at least 6 month

Exclusion Criteria:

* other condition that cause erectile dysfunction such as depression, hypogonadism, surgery, trauma, major cardiovascular event

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
clinical response to vardenafil | four weeks
  SEP 2; SEP 3 and IIEF variation

SECONDARY OUTCOMES:
endothelial dysfunction | four weeks
  variation of FMD of brachial artery from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Mario F Neves, MD, PhD., Study Chair — Hospital Universitario Pedro Ernesto; Valter Javaroni, MD, MSc, Principal Investigator — State University of Rio de Janeiro; Wille Oigman, MD, PhD, Study Director — State University of Rio de Janeiro
Locations (1):
- Hospital Universitário Pedro Ernesto, Rio de Janeiro, Rio de Janeiro, Brazil